CLINICAL TRIAL: NCT00640393
Title: A Randomized Study Combining Etanercept and Short Courses of Narrow-Band UVB in Patients With Psoriasis Vulgaris
Brief Title: Safety and Efficacy of Combining nbUVB to Etanercept in Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Inno-6007
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Results first posted 2010-12-14 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Psoriasis Vulgaris
Keywords: Etanercept, UVB, Enbrel, Psoriasis.
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 - Etanercept (Active Comparator): All participants received etanercept 50 mg twice a week for 12 weeks.
  Interventions: Drug: Etanercept
- Part 2 - Etanercept and nbUVB (Active Comparator): Participants who did not reach a 90 percent reduction in psoriasis area and severity index (PASI-90) after 12 weeks and were randomized to the narrow band ultra violet B (nbUVB) group. They received nbUVB treatments three times a week and 50 mg Etanercept once per week.
  Interventions: Drug: Etanercept; Device: nbUVB
- Part 2 - Etanercept (Active Comparator): Participants who did not reach PASI-90 after 12 weeks and were randomized to the Etanercept group. They received 50 mg Etanercept once per a week.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept 50 mg, subcutaneous (SC) injection.
  Other Names: Enbrel
Device: nbUVB
  Other Names: narrow band ultra violet B phototherapy; narrow band UVB
  Arms: Part 2 - Etanercept and nbUVB

SUMMARY:
This study will provide data on the addition of narrow band ultra violet B (nbUVB) phototherapy to participants who have not shown an excellent response to three months of etanercept.

DETAILED DESCRIPTION:
All participants will receive etanercept 50 mg twice a week for 12 weeks. Participants who reach PASI-90 at Day 84 will be discontinued from the study (they can continue receiving commercial etanercept outside the study). Participants remaining in the study at Day 84 will decrease etanercept to 50 mg weekly for another 12 weeks.

Participants who do not attain a 90 percent reduction in PASI from baseline (PASI-90) after 12 weeks will be randomized (1:1) to receive either etanercept alone or etanercept with short courses of narrow band ultra violet B (nbUVB)phototherapy. Participants randomized to the nbUVB group will receive nbUVB treatments three times a weeks for at least four weeks. At every planned study visit after Day 84, nbUVB treatment will be discontinued in participants who reach PASI-90. nbUVB phototherapy will be re-initiated for another four weeks at the subsequent planned study visit if they lose their PASI-90 response.

Efficacy will be evaluated with PASI, BSA and PGA by a blinded evaluator at Days 0, 28, 84, 112, 140 and 168. The effect of the treatment on quality of life will be evaluated using the DLQI questionnaire at Days 112, 140 and 168. Safety will be evaluated by physical examination and adverse events evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older;
* Patient with moderate to severe plaque psoriasis for whom a decision to use etanercept has been made;
* At the investigator discretion, patient who would benefit from systemic therapy;
* PASI (psoriasis area and severity index) ≥ 10 and BSA (body surface area affected by psoriasis) ≥ 10 at day 0;
* Unless surgically sterile (or at least 1 year post-menopausal for women), abstinent or homosexual, patient (men and women) willing to use adequate contraceptive method for at least 30 days before Day 0 and until one month after the last drug administration;
* Patient capable of giving informed consent;
* Patient with normal or non clinically significant chest X ray within six months of screening;
* Patient with negative purified protein derivative (PPD) within 3 months of Day 0;
* Negative urine pregnancy test for women of childbearing potential

Exclusion Criteria:

* Patient used topical steroid, topical tar preparations, or other anti-psoriatic preparations except tar or salicylic acid shampoo or hydrocortisone for the face, scalp, genital and inframammary areas within two weeks of Day 0;
* Patient with presence of erythrodermic, pustular or a predominantly guttate psoriasis;
* At the investigator's discretion, patient with any significant infection within 30 days of screening or a patient at risk of septicemia;
* Patient with evidence of any skin condition that would interfere with the evaluation of psoriasis;
* Patient used investigational drugs within 12 weeks or three half-life of Day 0 whichever is longer;
* Patient used systemic anti-psoriatic drugs such as steroids, retinoids, methotrexate, cyclosporine within four weeks of Day 0;
* Patient used any biologic such as alefacept, etanercept, efalizumab, infliximab and adalimumab within 12 weeks of Day 0;
* Patient used ultraviolet light therapy (UVB or nbUVB) within four weeks of Day 0 or PUVA (psoralen ultra violet A) within eight weeks of Day 0;
* Patient with prior or concurrent use of cyclophosphamide;
* Patient with concurrent sulfasalazine therapy or concurrent use of anakinra;
* Patient with an unstable or serious medical condition as defined by the investigator or presence of any significant medical condition that might cause this study to be detrimental to the patient.
* Uncontrolled or severe comorbidities such as diabetes mellitus requiring insulin; congestive heart failure (NYHA (New York Heart Association) class III or IV) or history of myocardial infarction or cerebrovascular accident or transient ischemic attack within three months of screening visit; unstable angina pectoris; uncontrolled hypertension, oxygen-dependent severe pulmonary disease;
* Patient with a known sero-positivity for HIV (human immunodeficiency virus) or history of any other immunosuppressing disease;
* Patient with active or chronic hepatitis B or C;
* Patient with any active or chronic infection within four weeks before screening or between the screening and baseline visits;
* Patient with any mycobacterial disease, patient with a positive PPD, a chest X-Ray suggestive of tuberculosis or patient taking anti-tuberculosis medication;
* Patient with a known hypersensitivity to etanercept or one of its components or known to have antibodies to etanercept;
* Patient who received a live attenuated vaccines within 12 weeks of Day 0 or plan to receive one during the study;
* Current pregnancy or lactation;
* At the investigator's discretion, patient with current or history of alcohol or drug abuse that would interfere with the ability of the patient to comply with the study protocol;
* Patient with systemic lupus erythematosus or demyelinating disorder (optic neuritis, multiple sclerosis or other);
* Patient with a history of cancer within five years of Day 0 or presence of cancer except for treated basal or squamous cell carcinoma and in situ cervix carcinoma;
* Patient who failed to respond to nbUVB in the past;
* Patient who have a contra-indication to nbUVB;
* Patient with latex sensitivity (applicable only if they are using prefilled syringe or prefilled SureClickTM autoinjector presentations);
* Patient with a history of non-compliance with other therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-04; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (10):
- Canada (10):
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Sudbury Skin Clinic, Greater Sudbury, Ontario
  - Mediprobe Research inc., London, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Bank on Beauty, Niagara Falls, Ontario
  - Innovaderm Research Laval Inc, Laval, Quebec
  - Clinique Dermatologique Fleury, Montreal, Quebec
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec Metropolitain, Québec, Quebec

REFERENCES:
- [Derived] Lynde CW, Gupta AK, Guenther L, Poulin Y, Levesque A, Bissonnette R. A randomized study comparing the combination of nbUVB and etanercept to etanercept monotherapy in patients with psoriasis who do not exhibit an excellent response after 12 weeks of etanercept. J Dermatolog Treat. 2012 Aug;23(4):261-7. doi: 10.3109/09546634.2011.607795. Epub 2011 Aug 10. PMID 21797805

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 2 - Etanercept and nbUVB: Participants who did not reach PASI-90 after 12 weeks and were randomized to the nbUVB group. They received nbUVB treatments three times a week and 50 mg Etanercept once per week.
- Part 2 - Etanercept: Participants who did not reach PASI-90 after 12 weeks were randomized to the Entercept group. They received 50 mg Etanercept once per a week.
Period: Part 1
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Started | 99 | 0 | 0
Completed | 94 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Period: Randomization
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Started | 94 | 0 | 0
Completed | 75 | 0 | 0
Not Completed | 19 | 0 | 0
Not completed — Withdrawn per protocol | 17 | 0 | 0
Not completed — Never randomized by site | 2 | 0 | 0
Period: Part 2
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Started | 0 | 37 | 38
Completed | 0 | 27 (Per Protocol analysis is of 7 participants that were compliant to protocol) | 35 (Per protocol analysis of 27 to 29 participants that were compliant depending on evaluation or visit)
Not Completed | 0 | 10 | 3
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 6 | 1
Not completed — Non-adherence | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Part 1 - Etanercept
Number analyzed (Participants) | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 94
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 43.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 68
Region of Enrollment [Number; unit: participants]
  Canada | 99
PASI - (Psoriasis area and severity index) [Mean (Standard Deviation); unit: Total units on a scale] — Four anatomic sites (head, upper extremities, trunk and lower extremities) are assessed for erythema, induration (plaque thickness), and desquamation (scaling) as seen on the day of the examination. The severity of each sign is assessed using a 5-point scale
  * 0 = No symptoms
  * 1 = Slight
  * 2 = Moderate
  * 3 = Marked
  * 4 = Very marked
  The area affected by psoriasis within a given anatomic site is estimated as a percentage of the total area of that anatomic site and assigned a numerical value according to the degree of psoriatic involvement from 0-6 Total scale 0 = best and 72 = worst
  Total units on a scale | 17.1 (7.4)
PGA - Physician's Global Assessment. [Mean (Standard Deviation); unit: Units on a scale] — The degree of overall lesion severity at the time of the physician's evaluation of the patient evaluated using the following scale:
  * 0 = clear
  * 1 = minimal
  * 2 = mild
  * 3 = moderate
  * 4 = severe
  * 5 = very severe
  The scale evaluates plaque elevation, scaling and erythema.
  Units on a scale | 3.6 (0.7)
BSA - Body surface area [Mean (Standard Deviation); unit: Percentage of the body affected] — Percentage of the body affected by psoriasis.
  Percentage of the body affected | 21.7 (14.2)
DLQI - Dermatology life quality index [Mean (Standard Deviation); unit: Units on a scale] — The aim of this questionnaire is to measure how much one's skin problem has affected one's life over the week prior to the visit.
  Scale is from 0 best to 30 worst.
  Units on a scale | 12.9 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Attaining a 90 Percent Reduction in PASI From Baseline (PASI 90) - ITT
Description: Four anatomic sites - head, upper extremities, trunk and lower extremities - are assessed for erythema, induration, and desquamation. The severity of each sign is assessed using a 5-point scale:
  * 0 = No symptoms
  * 1 = Slight
  * 2 = Moderate
  * 3 = Marked
  * 4 = Very marked
  The area affected by psoriasis within a given anatomic site is estimated as a percentage of the total area of that anatomic site and assigned a numerical value according to the degree of psoriatic involvement from 0-6.
  Total scale 0 = best and 72 = worst
Time Frame: 112 and 140 days
Population: The analysis was intention to treat (ITT) and the imputation technique was Non-Responder(NRI).
Measure: Number; unit: Participants
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 0 | 37 | 38
Participants
  Day 84 |  | 0 | 0
  Day 112 |  | 3 | 1
  Day 140 |  | 5 | 5
  Day 168 |  | 6 | 6

2. Secondary Outcome: Number of Participants Attaining a 75 Percent Reduction in PASI From Baseline (PASI 75) - ITT
Description: as for outcome 1
Time Frame: 112, 140 and 168 days
Population: The analysis was intention to treat (ITT) and the imputation technique was Non-Responder(NRI).
Measure: Number; unit: Participants
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 0 | 37 | 38
Participants
  Day 84 |  | 18 | 13
  Day 112 |  | 15 | 12
  Day 140 |  | 23 | 17
  Day 168 |  | 19 | 17

3. Secondary Outcome: Number of Participants Attaining a 100% Reduction in PASI From Baseline (PASI 100) - ITT
Description: as for outcome 1
Time Frame: 112, 140 and 168 days
Population: The analysis was intention to treat (ITT) and the imputation technique was Non-Responder (NRI).
Measure: Number; unit: Participants
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 0 | 37 | 38
Participants
  Day 84 |  | 0 | 0
  Day 112 |  | 2 | 0
  Day 140 |  | 1 | 1
  Day 168 |  | 2 | 2

4. Secondary Outcome: Number of Participants Attaining a 50% Reduction From Baseline in PASI From Baseline (PASI-50) - ITT
Description: as for outcome 1
Time Frame: 28 and 84 days
Population: The analysis was intention to treat (ITT) and the imputation technique was Non-Responder (NRI).
Measure: Number; unit: Participants
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 99 | 0 | 0
Participants
  Day 28 | 37 |  |
  Day 84 | 82 |  |

5. Secondary Outcome: Number of Participants Attaining a 75 % Reduction in PASI From Baseline (PASI-75) - ITT
Description: as for outcome 1
Time Frame: 28 and 84 days
Population: The analysis was intention to treat (ITT) and the imputation technique was Non-Responder (NRI).
Measure: Number; unit: Participants
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 99 | 0 | 0
Participants
  Day 28 | 13 |  |
  Day 84 | 50 |  |

6. Secondary Outcome: Number of Participants Attaining a 90 Percent Reduction in PASI From Baseline (PASI-90) - ITT
Description: as for outcome 1
Time Frame: 28 and 84 days
Population: The analysis was intention to treat (ITT) and the imputation technique was Non-Responder (NRI).
Measure: Number; unit: Participants
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 99 | 0 | 0
Participants
  Day 28 | 3 |  |
  Day 84 | 17 |  |

7. Secondary Outcome: Number of Participants Attaining a 100 Percent Reduction in PASI From Baseline (PASI-100) - ITT
Description: as for outcome 1
Time Frame: 28 and 84 days
Population: The analysis was intention to treat (ITT) and the imputation technique was Non-Responder (NRI).
Measure: Number; unit: Participants
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 99 | 0 | 0
Participants
  Day 28 | 2 |  |
  Day 84 | 8 |  |

8. Secondary Outcome: Number of Patients Attaining a PGA (Physician's Global Assessment) of 0 or 1 - ITT
Description: Number of patients attaining a Physician's Global Assessment (PGA) of clear (0) or minimal (1).
  PGA scores are evaluated at each time point.
  The degree of overall lesion severity at the time of the physician's evaluation of the patient evaluated using the following scale:
  * 0 = clear
  * 1 = minimal
  * 2 = mild
  * 3 = moderate
  * 4 = severe
  * 5 = very severe
  The scale evaluates plaque elevation, scaling and erythema.
Time Frame: 0, 112, 140 and 168 days
Population: The analysis was intention to treat (ITT) and the imputation technique was Non Responder (NRI).
Measure: Number; unit: Participants
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 0 | 37 | 38
Participants
  Day 84 |  | 11 (0.6) | 11 (0.72)
  Day 112 |  | 13 (0.88) | 8 (0.88)
  Day 140 |  | 13 (0.79) | 11 (0.94)
  Day 168 |  | 12 (0.86) | 13 (1.01)

9. Secondary Outcome: Body Surface Area (BSA) Affected by Psoriasis - ITT
Description: BSA scores are evaluated at each time point.
  BSA is a measure of the percentage of body surface affected by psoriasis.
Time Frame: 0, 84, 112, 140 and 168 days
Population: The analysis was intention to treat (ITT) and the imputation technique was Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Percent of body affected
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 0 | 37 | 38
Percent of body affected
  Day 0 |  | 19.06 (12.68) | 23.65 (16.91)
  Day 84 |  | 6.69 (6.95) | 8.28 (7.98)
  Day 112 |  | 4.92 (5.38) | 7.27 (7.16)
  Day 140 |  | 4.43 (5.57) | 6.53 (7.73)
  Day 168 |  | 3.28 (2.58) | 7.19 (8.17)

10. Secondary Outcome: Dermatology Life Quality Index (DLQI) - ITT
Description: The aim of this questionnaire is to measure how much one's skin problem has affected one's life over the week prior to the visit.
  Questionnaire is patient-assessed (self-reported). DLQI scores are evaluated at each time point.
  Scale is from 0 best to 30 worst.
  0-1 = no effect at all on patient's life 2-5 = small effect on patient's life 6-10 = moderate effect on patient's life 11-20 = very large effect on patient's life 21-30 = extremely large effect on patient's life
Time Frame: 0, 84, 112, 140 and 168 days
Population: The analysis was intention to treat (ITT) and the imputation technique was Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 0 | 37 | 38
Units on a scale
  Day 0 |  | 11.92 (6.49) | 12.47 (6.93)
  Day 84 |  | 3.69 (3.36) | 5.97 (6.28)
  Day 112 |  | 3.06 (3.23) | 6.03 (5.57)
  Day 140 |  | 2.69 (2.86) | 6.05 (5.87)
  Day 168 |  | 2.83 (3.26) | 6.00 (6.07)

11. Secondary Outcome: Number of Adverse Drug Reactions - ITT
Description: Evaluation of safety of etanercept and nbUVB as compared to etanercept alone by reporting the incidence rates of adverse drug reactions.
  Definition: A response to a drug that is noxious and unintended and that occurs at doses normally used in man for prophylaxis, diagnosis, or therapy of diseases or for modification of physiological function.
  Only adverse drug reactions that were at least possibly related to etanercept were recorded. All symptoms observed at the injection site such as erythema, burning, edema and pruritus were recorded together as Injection Site Reaction.
Time Frame: 196 days
Population: The analysis was intention to treat (ITT).
Measure: Number; unit: Adverse drug reactions.
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 99 | 37 | 38
Adverse drug reactions. | 7 | 3 | 2

12. Secondary Outcome: Number of Infectious Adverse Events - ITT
Description: Evaluation of safety of etanercept and nbUVB as compared to etanercept alone by reporting the incidence rates of infectious adverse events.
  Definition: An adverse event is any untoward medical occurrence in a patient administered a pharmaceutical product, without regard to the possibility of a causal relationship with this treatment.
  Only infectious and malignant (including any type of skin cancer) adverse events were recorded.
Time Frame: 196 days
Population: The analysis was intention to treat (ITT).
Measure: Number; unit: Infectious adverse events
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 99 | 37 | 38
Infectious adverse events | 21 | 7 | 17

13. Secondary Outcome: Number of Serious Adverse Events - ITT
Description: Evaluation of safety of etanercept and nbUVB as compared to etanercept alone by reporting the incidence rates of serious adverse events.
  Definition: any adverse event from this study that results in one of the following outcomes, or is significant for any other reason:
  * death
  * initial or prolonged inpatient hospitalization
  * a life-threatening experience (that is, immediate risk of dying)
  * persistent or significant disability/incapacity
  * congenital anomaly/birth defect
Time Frame: 196 days
Population: The analysis was intention to treat (ITT).
Measure: Number; unit: Serious adverse events
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 99 | 37 | 38
Serious adverse events | 1 | 0 | 2

14. Secondary Outcome: Number of Participants Attaining a 90 Percent Reduction in PASI From Baseline (PASI 90) - PP
Description: as for outcome 1
Time Frame: 84, 112, 140 and 168 days
Population: The analysis was per protocol (PP). Participants that were not 80 percent compliant to narrow band UVB treatment at each visit and patients that missed excessive etanercept injections were excluded completely from analysis. One patient missed a visit at Day 140 but was compliant to protocol.
Measure: Number; unit: Participants
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 0 | 7 | 29
Participants
  Day 84 |  | 0 | 0
  Day 112 |  | 3 | 1
  Day 140 (n = 28 for etanercept) |  | 3 | 5
  Day 168 |  | 3 | 6

15. Secondary Outcome: Number of Participants Attaining a 75 Percent Reductionin PASI From Baseline (PASI-75) - PP
Description: as for outcome 1
Time Frame: 84, 112, 140 and 168 days
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 0 | 7 | 29
Participants
  Day 84 |  | 3 | 11
  Day 112 |  | 6 | 12
  Day 140 (n = 28 for etanercept) |  | 7 | 16
  Day 168 |  | 7 | 16

16. Secondary Outcome: Number of Participants Attaining a 100 Percent Reduction in PASI From Baseline (PASI-100) - PP
Description: as for outcome 1
Time Frame: 84, 112, 140 and 168 days
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 0 | 7 | 29
Participants
  Day 84 |  | 0 | 0
  Day 112 |  | 2 | 0
  Day 140 (n = 28 for etanercept) |  | 1 | 1
  Day 168 |  | 1 | 2

17. Secondary Outcome: Number of Patients Attaining a PGA (Physician's Global Assessment) of 0 or 1 - PP
Description: as for outcome 8
Time Frame: 84, 112, 140 and 168 days
Population: The analysis was per protocol (PP). Participants that were not 80 percent compliant to narrow band UVB treatment at each visit and patients that missed excessive etanercept injections were excluded completely from analysis. One patient missed a visit at Day 140 but was compliant to protocol. And PGA was not performed for another patient (Day 168)
Measure: Number; unit: Participants
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 0 | 7 | 29
Participants
  Day 84 |  | 4 (0.49) | 9 (0.69)
  Day 112 |  | 5 (0.82) | 6 (0.97)
  Day 140 (n = 28 for etanercept) |  | 6 (0.58) | 9 (1.05)
  Day 168 (n = 28 for etanercept) |  | 7 (0.38) | 11 (1.05)

18. Secondary Outcome: Body Surface Area (BSA) Affected by Psoriasis - PP
Description: BSA scores are evaluated at each time point.
  BSA is a measure of the percentage of body surface affected by psoriasis.
Time Frame: 0, 84, 112, 140 and 168 days
Population: The analysis was per protocol (PP). Participants that were not 80 percent compliant to narrow band UVB treatment at each visit and patients that missed excessive etanercept injections were excluded completely from analysis. One patient missed a visit at Day 140.
Measure: Mean (Standard Deviation); unit: Percent of body affected
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 0 | 7 | 28
Percent of body affected
  Day 0 |  | 17.82 (8.72) | 24.24 (16.89)
  Day 84 |  | 6.04 (4.78) | 8.63 (8.67)
  Day 112 |  | 2.93 (4.97) | 7.57 (7.93)
  Day 140 |  | 2.07 (2.28) | 6.68 (8.69)
  Day 168 |  | 1.57 (1.54) | 7.21 (8.42)

19. Secondary Outcome: Dermatology Life Quality Index (DLQI) - PP
Description: as for outcome 10
Time Frame: 0, 84, 112, 140 and 168 days
Population: The analysis was per protocol (PP). Participants that were not 80 percent compliant to narrow band UVB treatment at each visit and patients that missed excessive etanercept injections were excluded completely from analysis. One patient missed a visit at Day 140. Results for one were excluded because of missing DLQI questionnaire results.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Number analyzed (Participants) | 0 | 7 | 27
Units on a scale
  Day 0 |  | 9.43 (6.24) | 12.3 (7.7)
  Day 84 |  | 3.00 (1.53) | 6.07 (5.98)
  Day 112 |  | 1.71 (1.89) | 5.89 (5.53)
  Day 140 |  | 0.71 (0.95) | 6.00 (6.08)
  Day 168 |  | 0.57 (0.79) | 5.89 (6.27)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 12 week period for part 1 and over a 16 week period for part 2.
Arm/Group | Part 1 - Etanercept | Part 2 - Etanercept and nbUVB | Part 2 - Etanercept
Serious Adverse Events (participants affected / at risk) | 1/99 | 0/37 | 2/38
Other Adverse Events (participants affected / at risk) | 17/99 | 3/37 | 11/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - Etanercept (N=99) | Part 2 - Etanercept and nbUVB (N=37) | Part 2 - Etanercept (N=38)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Low blood pressure (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - Etanercept (N=99) | Part 2 - Etanercept and nbUVB (N=37) | Part 2 - Etanercept (N=38)
Common cold (Infections and infestations) | 9 (9) | 2 (2) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 6 (6)
Injection site reaction (General disorders) | 4 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less